CLINICAL TRIAL: NCT03865602
Title: Improving Morbidity During Post-Acute Care Transitions for Sepsis (IMPACTS): A Pragmatic Randomized Evaluation of Implementing Best Practice Care for Sepsis Survivors to Reduce Morbidity and Mortality
Brief Title: Improving Morbidity During Post-Acute Care Transitions for Sepsis
Acronym: IMPACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00082326; 01-19-24E (Other: Atrium)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Clinical Sepsis
Keywords: evidence based medicine; continuity of patient care; patient navigator; health services; pragmatic clinical trial
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sepsis Transition And Recovery (STAR) (Experimental): Virtual sepsis navigation delivered across the peri-hospital discharge interval
  Interventions: Behavioral: Sepsis Transition And Recovery (STAR)
- Usual Care (Active Comparator): Patients and their providers will have no access to the STAR program. Aspects of usual care will be determined by treating clinicians independent of trial assignment.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Sepsis Transition And Recovery (STAR) — In the STAR program intervention, a centrally located nurse navigator facilitates the application of four evidence-based core components of post-sepsis care (i.e., review of medications, new impairments, comorbidities, and palliative care) to patients prior to and during the 30 days after hospital discharge. The STAR navigator will provide telephone and EHR-based support within the hospitalization and to patients across all discharge settings with remote monitoring at specified intervals following hospital discharge. Patients will continue to receive STAR directed services for 30 days following their discharge and then will be transitioned back to the next appropriate care location.
  Arms: Sepsis Transition And Recovery (STAR)
Behavioral: Usual care — Patients and their providers will not have access to the STAR program. Patients will continue to receive usual care throughout their stay and discharge, consisting of: patient education and follow-up instructions at discharge, which are not specific to sepsis; routine recommendations for follow-up visits with primary care providers; arrangements for home health services or care management follow-up based on each patient's needs but not specifically tailored to the sepsis population; discharge to post-acute setting with no sepsis-specific follow-up. All aspects of usual care will be determined by treating clinicians independent of trial assignment.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to improve transitions of care for the highest risk, complex patients with suspected sepsis. Atrium Health has developed a nurse-navigator facilitated care transition strategy, called the Sepsis Transition and Recovery (STAR) program, to improve the implementation of recommended care practices and bridge care gaps for patients in the post-sepsis transition period. During their hospitalization, STAR program patients enter into a transition pathway facilitated by a centrally located nurse navigator and including the following evidence-based post-sepsis care components: i) review and recommendation for adjustment of medications; ii) identification of and referral for new physical, mental, and cognitive deficits; iii) surveillance for treatable conditions that commonly lead to poor outcomes; and iv) referral to palliative care when appropriate. IMPACTS (Improving Morbidity during Post-Acute Care Transitions for Sepsis) is a pragmatic, randomized program evaluation to compare clinical outcomes between sepsis survivors who receive usual care versus care delivered through the STAR program following hospitalization. IMPACTS will test the hypothesis that patients that receive care through STAR will have decreased composite all cause, 30-day hospital readmission and mortality compared to patients that receive usual care.

DETAILED DESCRIPTION:
BACKGROUND

Sepsis is a common and life-threatening condition defined by organ dysfunction due to a dysregulated response to infection (Fleischmann, 2016). Aggressive early sepsis identification and treatment initiatives have decreased hospital mortality for patients with sepsis (Rhodes, 2017). As mortality rates have improved, there has been a growing recognition of the downstream effects of sepsis for the approximately 14 million annual sepsis survivors who encounter increased long-term mortality and morbidity across functional, cognitive, and psychological domains (Iwashyna, 2010; Shah, 2013; Schuler, 2018; Borges, 2015; Annane, 2015; Prescott, 2015). Currently, there is a disconnect between the post-acute care needs of sepsis survivors and the resources available to these patients (Huang, 2016; Ortego, 2015; Winters, 2010; Nesseler, 2013). Inadequate post-sepsis care strategies are reflected by adverse outcomes post-sepsis including increased mortality risk and strikingly high rates of healthcare utilization, including a 90-day hospital readmission rate of 40% and over 3 billion dollars in preventable costs (Prescott, 2016; Goodwin, 2015; Prescott, 2014; Jones, 2015). To address the specific gaps in treatment for sepsis survivors, international experts developed best-practice recommendations to guide delivery of post-sepsis care (Prescott, 2018). These best-practice recommendations are directed towards the specific challenges and sequelae following a sepsis hospitalization and include: i) identification and treatment of new physical, mental, and cognitive deficits; ii) review and adjustment of medications; iii) surveillance of treatable conditions that commonly lead to poor outcomes; and iv) focus on palliative care when appropriate. However, implementation of recommended post-sepsis practices is hindered by a gap in understanding how to best integrate interventions into the complex and fragmented post discharge setting (e.g., lack of provider time and patient engagement, limited access to care management, and insufficient institutional support) (Taylor, 2019; Brownson, 2012; Bodenheimer, 2008; Coleman, 2004).

RATIONALE

In randomized controlled trials (RCTs), including our previous work, successfully implemented care transition programs using nurse navigators have been shown to reduce hospital readmissions and costs. To better enhance transitions of care for the highest risk, complex patients with suspected sepsis, we propose extending this evidence using a nurse-facilitated care transition program for patients in the post-sepsis transition period to improve the implementation of recommended care practices and bridge care gaps. This approach, called the Sepsis Transition and Recovery (STAR) program, is the next step in the progression of our group's work on improving discharge transitions and sepsis processes of care. A key aspect of this initiative includes the ability to identify sepsis survivors at the greatest risk for poor outcomes. For example, one-quarter of sepsis survivors account for three-quarters of hospital readmissions and costs, indicating that identifying high-risk sepsis patients for targeted facilitation of best-practice care could efficiently impact quality and cost.

Our STAR program uses near real-time risk modeling to identify high-risk patients and a centrally located nurse, virtually connected to participating hospitals, to coordinate the application of evidence-based recommendations for post-sepsis care, overcome barriers to recommended care, and bridge gaps in service that can serve as points of failure for complex patients. During their hospitalization, high-risk patients enter into a transition pathway integrated within Atrium Health Hospital Medicine's Transition Services program and includes the following core components: i) Introduction to STAR process prior to discharge (confirm provider consults e.g., PT, ID, palliative); ii) Disease-specific education and discharge "playbook"; iii) Virtual hospital follow-up evaluation within 48 hours including medication reconciliation; iv) Second, post-acute virtual follow-up within 72 hours (symptom monitoring, confirm provider follow-up); v) Weekly contact with care management team; vi) Referral to provider follow-up (e.g., primary care provider, transition clinic) as appropriate; vii) Coordinated transition to the next appropriate care location after 30 days from time of discharge. The STAR navigator also meets weekly with the Medical Director of the Atrium Health Transition Services program who provides additional clinical oversight of ongoing cases.

The IMPACTS (Improving Morbidity during Post Acute Care Transitions for Sepsis) evaluation will examine if implementation of the STAR program within a large healthcare system will improve outcomes for high-risk sepsis patients. This randomized program evaluation is designed to be a seamless part of routine care in a real-world setting to generate knowledge of best practices for implementation and dissemination of post-sepsis transitions of care.

INVESTIGATIONAL PLAN

Overall Study Design

This real-world pragmatic randomized program evaluation will compare the effectiveness of the Sepsis Transition And Recovery (STAR) program versus usual care on post-sepsis care and patient outcomes. The STAR program is informed by existing evidence and designed using the Chronic Care Model to increase best-practice adherence and care coordination, resulting in improved transitions between hospitals and post-acute care during sepsis recovery.

Because of resource limitations, STAR can only be made available to a limited number of patients. To be objective in patient selection and allow for program evaluation, we will use a data driven approach to identify patients as eligible for program referral. First, risk modeling will identify patients as high risk for 30-day readmission or 30-day mortality during the first day of the hospital admission. Then from this pool of high-risk patients, up to 6 patients will be randomly selected each weekday to be referred to either receive usual care or care delivered through the STAR program. The number of daily patients to be randomized was selected to match targeted capacity for the STAR navigator and will be reevaluated on a biweekly basis. Because variables that affect eligibility may change during a hospital stay, initial eligibility will be re-confirmed at time of hospital discharge. Specifically, patients who have had infection diagnosis ruled-out during their hospitalization (i.e., rule-out documented in medical record) will be excluded for the purposes of analysis. All remaining eligible patients at the time of discharge will be included in analyses, which will be conducted using an intent-to-treat approach. Planned enrollment is 708 patients (n=354 patients per study arm) and STAR program follow-up will be completed 30 days after hospital discharge. Outcomes data will be tracked for 90 days and captured from routinely collected data from the Atrium Health Enterprise Data Warehouse. Given this evaluation protocol is part of a quality improvement intervention that relies on using evidence-based interventions, only utilizes data collected as part of routine care, and is minimal risk to patients, we requested that the institutional review board designate this study as expedited research and grant a waiver of informed consent.

Primary Outcome Variable The primary outcome is a composite, dichotomous endpoint of all-cause mortality or unplanned hospital readmission assessed 30 days post index hospital discharge.

Secondary Outcome Variable(s)

1. all-cause 30- and 90-day mortality;
2. all-cause 30- and 90-day hospital readmission;
3. 30- and 90-day cause-specific hospital readmissions with primary diagnoses related to: a) infection, b) chronic lung disease, c) heart failure, and d) acute kidney injury;
4. 30- and 90-day emergency department visits;
5. 30- and 90-day acute-care costs;
6. 30- and 90-day total healthcare costs (only in the subgroup of patients enrolled in a Medicare Shared Savings Plan);
7. acute care-free days alive measured at 30 and 90 days, defined as the sum of days alive without inpatient, observation, and emergency department encounters (rounded to full day for any day with acute care utilization) during the interval after discharge.

Subject Selection Subject selection will occur via an automated query process for patient list generation. Each weekday morning actively admitted patients at 3 study hospitals (i.e., Carolinas Medical Center, Carolinas Medical Center - Mercy, and Atrium Health Northeast) will be identified from the electronic health record and Enterprise Data Warehouse and output into daily eligibility lists based on the study's inclusion/exclusion criteria.

Randomization Eligible patients will be randomly allocated 1:1 to receive usual care or the STAR program. Clinicians and patients are not blinded to treatment allocation. Due to resource limitations, STAR will only be made available to a limited number of patients. Thus, a constrained randomization scheme will be utilized to randomly allocate up to six eligible patients to either STAR or usual care each weekday. The number of patients allocated to be randomized daily was selected to match targeted capacity for the STAR navigators and will be reevaluated on a biweekly basis and adjusted as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted from the emergency department to inpatient or observation status at one of: Carolinas Medical Center, Carolinas Medical Center - Mercy, or Atrium Health Northeast;
2. ≥18 years of age upon admission;
3. oral/parenteral antibiotic or bacterial culture order within 24 hours of emergency department presentation and

   1. culture drawn first, antibiotics ordered within 48 hours or
   2. antibiotics ordered first, culture ordered within 48 hours (adapted from criteria applied in development of the Third International Consensus Definitions for Sepsis and Septic Shock)
4. deemed as high-risk for 30-day readmission (i.e., ≥ 20%) or 30-day mortality (i.e., ≥ 10%) using risk-scoring models
5. not discharged at the time of patient list generation

Exclusion Criteria:

1. prior randomization to either STAR or usual care study arms;
2. not a North Carolina resident or residence >2.5-hour drive time from treating hospital;
3. the only antibiotic associated with patient is administered in the operating room as this likely represents pre-operative infection prophylaxis and not presumed infection;
4. patients transferred from other acute care hospitals;
5. patients with a change in code status (i.e., do not resuscitate, do not intubate) within 24 hours after admission due to the general assumption of increased risk of exposure to less aggressive treatment;
6. patients with infection ruled out during the index hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Combined all-cause mortality or unplanned hospital readmission | 30 days from index visit
  Hospital readmission will be captured from healthcare utilization data in the Atrium Health enterprise data warehouse. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility. Vital status verification data is ascertained via monthly Social Security Administration Limited Access Death Master File (DMF) data feed and validated record linkage process into the Atrium Health data warehouse. For the composite primary outcome, we will capture all patients with either date of death or eligible hospital readmission prior to 30 days post discharge as event-positive.

SECONDARY OUTCOMES:
All-cause mortality | 30 days from index visit
  Death inside or outside of the hospital ascertained via monthly Social Security Administration Limited Access Death Master File (DMF) data feed and validated record linkage process into the Atrium Health data warehouse.
All-cause mortality | 90 days from index visit
  Death inside or outside of the hospital ascertained via monthly Social Security Administration Limited Access Death Master File (DMF) data feed and validated record linkage process into the Atrium Health data warehouse.
All-cause unplanned hospital readmission | 30 days from index visit
  Hospital readmission will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
All-cause unplanned hospital readmission | 90 days from index visit
  Hospital readmission will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Infection-related unplanned hospital readmission | 30 days from index visit
  Hospital readmission with infection-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Infection-related unplanned hospital readmission | 90 days from index visit
  Hospital readmission with infection-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Chronic lung disease-related unplanned hospital readmission | 30 days from index visit
  Hospital readmission with chronic lung disease-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Chronic lung disease-related unplanned hospital readmission | 90 days from index visit
  Hospital readmission with chronic lung disease-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Heart failure-related unplanned hospital readmission | 30 days from index visit
  Hospital readmission with heart failure-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Heart failure-related unplanned hospital readmission | 90 days from index visit
  Hospital readmission with heart failure-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Acute kidney injury-related unplanned hospital readmission | 30 days from index visit
  Hospital readmission with acute kidney injury-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
Acute kidney injury-related unplanned hospital readmission | 90 days from index visit
  Hospital readmission with acute kidney injury-related primary discharge diagnosis will be captured from any Atrium Health facility. Index visit is defined by the Centers for Medicaid and Medicare Services (CMS) with additional inclusion of observation patients at any Atrium Health facility.
All-cause emergency department visits | 30 days from index visit
  Emergency department visits to any Atrium Health facility
All-cause emergency department visits | 90 days from index visit
  Emergency department visits to any Atrium Health facility
Acute care costs | 30 days from index visit
  Costs attributed to acute care received at any Atrium Health emergency department, observation, or inpatient hospital encounter
Acute care costs | 90 days from index visit
  Costs attributed to acute care received at any Atrium Health emergency department, observation, or inpatient hospital encounter
Total healthcare costs | 30 days from index visit
  Costs attributed to healthcare claims incurred at any Atrium Health or outside system facility (only in the subgroup of patients enrolled in a Medicare Shared Savings Plan)
Total healthcare costs | 90 days from index visit
  Costs attributed to healthcare claims incurred at any Atrium Health or outside system facility (only in the subgroup of patients enrolled in a Medicare Shared Savings Plan)
Acute care-free days alive | 30 days from index visit
  The sum of days alive without inpatient, observation, and emergency department encounters at any Atrium Health facility (rounded to full day for any day with acute care utilization) during the interval after discharge
Acute care-free days alive | 90 days from index visit
  The sum of days alive without inpatient, observation, and emergency department encounters at any Atrium Health facility (rounded to full day for any day with acute care utilization) during the interval after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kowalkowski, PhD, Principal Investigator — Wake Forest University Health Sciences; Stephanie P Taylor, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Shah FA, Pike F, Alvarez K, Angus D, Newman AB, Lopez O, Tate J, Kapur V, Wilsdon A, Krishnan JA, Hansel N, Au D, Avdalovic M, Fan VS, Barr RG, Yende S. Bidirectional relationship between cognitive function and pneumonia. Am J Respir Crit Care Med. 2013 Sep 1;188(5):586-92. doi: 10.1164/rccm.201212-2154OC. PMID 23848267
- [Background] Schuler A, Wulf DA, Lu Y, Iwashyna TJ, Escobar GJ, Shah NH, Liu VX. The Impact of Acute Organ Dysfunction on Long-Term Survival in Sepsis. Crit Care Med. 2018 Jun;46(6):843-849. doi: 10.1097/CCM.0000000000003023. PMID 29432349
- [Background] Borges RC, Carvalho CR, Colombo AS, da Silva Borges MP, Soriano FG. Physical activity, muscle strength, and exercise capacity 3 months after severe sepsis and septic shock. Intensive Care Med. 2015 Aug;41(8):1433-44. doi: 10.1007/s00134-015-3914-y. Epub 2015 Jun 25. PMID 26109398
- [Background] Annane D, Sharshar T. Cognitive decline after sepsis. Lancet Respir Med. 2015 Jan;3(1):61-9. doi: 10.1016/S2213-2600(14)70246-2. Epub 2014 Nov 28. PMID 25434614
- [Background] Prescott HC, Langa KM, Iwashyna TJ. Readmission diagnoses after hospitalization for severe sepsis and other acute medical conditions. JAMA. 2015 Mar 10;313(10):1055-7. doi: 10.1001/jama.2015.1410. No abstract available. PMID 25756444
- [Background] Huang C, Daniels R, Lembo A, et al. Sepsis survivors' satisfaction with support services during and after their hospitalization. Crit Care Med. 2016;44(12):425.
- [Background] Ortego A, Gaieski DF, Fuchs BD, Jones T, Halpern SD, Small DS, Sante SC, Drumheller B, Christie JD, Mikkelsen ME. Hospital-based acute care use in survivors of septic shock. Crit Care Med. 2015 Apr;43(4):729-37. doi: 10.1097/CCM.0000000000000693. PMID 25365724
- [Background] Winters BD, Eberlein M, Leung J, Needham DM, Pronovost PJ, Sevransky JE. Long-term mortality and quality of life in sepsis: a systematic review. Crit Care Med. 2010 May;38(5):1276-83. doi: 10.1097/CCM.0b013e3181d8cc1d. PMID 20308885
- [Background] Nesseler N, Defontaine A, Launey Y, Morcet J, Malledant Y, Seguin P. Long-term mortality and quality of life after septic shock: a follow-up observational study. Intensive Care Med. 2013 May;39(5):881-8. doi: 10.1007/s00134-013-2815-1. Epub 2013 Jan 29. PMID 23358541
- [Background] Prescott HC, Osterholzer JJ, Langa KM, Angus DC, Iwashyna TJ. Late mortality after sepsis: propensity matched cohort study. BMJ. 2016 May 17;353:i2375. doi: 10.1136/bmj.i2375. PMID 27189000
- [Background] Goodwin AJ, Rice DA, Simpson KN, Ford DW. Frequency, cost, and risk factors of readmissions among severe sepsis survivors. Crit Care Med. 2015 Apr;43(4):738-46. doi: 10.1097/CCM.0000000000000859. PMID 25746745
- [Background] Prescott HC, Langa KM, Liu V, Escobar GJ, Iwashyna TJ. Increased 1-year healthcare use in survivors of severe sepsis. Am J Respir Crit Care Med. 2014 Jul 1;190(1):62-9. doi: 10.1164/rccm.201403-0471OC. PMID 24872085
- [Background] Jones TK, Fuchs BD, Small DS, Halpern SD, Hanish A, Umscheid CA, Baillie CA, Kerlin MP, Gaieski DF, Mikkelsen ME. Post-Acute Care Use and Hospital Readmission after Sepsis. Ann Am Thorac Soc. 2015 Jun;12(6):904-13. doi: 10.1513/AnnalsATS.201411-504OC. PMID 25751120
- [Background] Prescott HC, Angus DC. Enhancing Recovery From Sepsis: A Review. JAMA. 2018 Jan 2;319(1):62-75. doi: 10.1001/jama.2017.17687. PMID 29297082
- [Background] Taylor S, Figueroa-Sierra M, Shuman T, et al. Post-sepsis care recommendations are associated with improved patient outcomes but adherence is low [abstract]. Critical Care Medicine. 2019;47(1):636.
- [Background] Brownson RC, Allen P, Duggan K, Stamatakis KA, Erwin PC. Fostering more-effective public health by identifying administrative evidence-based practices: a review of the literature. Am J Prev Med. 2012 Sep;43(3):309-19. doi: 10.1016/j.amepre.2012.06.006. PMID 22898125
- [Background] Bodenheimer T. Coordinating care--a perilous journey through the health care system. N Engl J Med. 2008 Mar 6;358(10):1064-71. doi: 10.1056/NEJMhpr0706165. No abstract available. PMID 18322289
- [Background] Coleman EA, Berenson RA. Lost in transition: challenges and opportunities for improving the quality of transitional care. Ann Intern Med. 2004 Oct 5;141(7):533-6. doi: 10.7326/0003-4819-141-7-200410050-00009. PMID 15466770
- [Derived] Dellinger RP, Levy MM, Schorr CA, Townsend SR. 50 Years of Sepsis Investigation/Enlightenment Among Adults-The Long and Winding Road. Crit Care Med. 2021 Oct 1;49(10):1606-1625. doi: 10.1097/CCM.0000000000005203. No abstract available. PMID 34342304
- [Derived] Kowalkowski M, Chou SH, McWilliams A, Lashley C, Murphy S, Rossman W, Papali A, Heffner A, Russo M, Burke L, Gibbs M, Taylor SP; Atrium Health ACORN Investigators. Structured, proactive care coordination versus usual care for Improving Morbidity during Post-Acute Care Transitions for Sepsis (IMPACTS): a pragmatic, randomized controlled trial. Trials. 2019 Nov 29;20(1):660. doi: 10.1186/s13063-019-3792-7. PMID 31783900